CLINICAL TRIAL: NCT02960334
Title: Screening for Actionable Atrial Fibrillation During Preoperative Consultation With the MyDiagnostick
Status: Completed | Type: Observational
Sponsor: Martini Hospital Groningen (Other)
Responsible Party: Principal Investigator, Eva Roseboom, Student, Martini Hospital Groningen
Other Study IDs: 2016-076
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
Keywords: Screening; Silent Atrial Fibrillation; Undertreated Atrial Fibrillation; Actionable Atrial Fibrillation; MyDiagnostick; Opportunistic Screening; Preoperative Consultation; OAC; VKA; NOAC
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: MyDiagnostick — The MyDiagnostick is a compact hand-held device that registers and stores I-lead ECG strips. In one minute, t analyses the rhythm for the presence of AF. It distinguishes AF from normal cardiac rhythms by measuring RR-irregularity.

SUMMARY:
Atrial Fibrillation (AF) It is the most common arrhythmia in the world. It carries great public health significance because of its prevalence, additional morbidity and mortality. It provides a 4-5 times higher risk of developing a ischemic stroke or transient ischemic attack. In term, this risk can be 70% reduced by taking oral anticoagulants. Actionable AF is the overarching term for silent AF (asymptomatic AF) and undertreated AF (known AF, but not sufficiently protected against ischemic stroke). It is recommended that over the age of 65, patients should be screened with pulse palpation or rhythm strip for the presence of AF. The MyDiagnostick is a single-lead I, compact hand-held device that analyses heart rhythm during one minute. During preoperative consultation, this device will be used to value the yield of screening for actionable AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia in the world, with a prevalence ranging from 1.9 - 2.3% and rising. It is known that the disease occurs more often as age progresses: 70% of affected cases are aged between 65 and 85, over 80 years, one is 10-18% likely to be carrying the illness. Multiple risk factors for developing AF have been determined, like hypertension, myocardial infarction, heart failure, valvular heart disease, obesity, DM and hyperthyroidism.

AF potentially leads to thrombus formation, resulting in a 4-5 times increased risk of getting a TIA or ischemic infarction.

Taking a 12 lead electrocardiogram (ECG) remains the golden standard, with the absence of distinct P-waves and a RR interval that is irregularly irregular.

AF is a risk factor and a risk marker for developing ischemic stroke, by providing a prothrombotic environment. This makes a patient with AF 4-5 times more susceptible for getting an ischemic stroke. Protection for this risk is done by prescribing oral anticoagulants (OAC) (according to an individuals CHA2DS2VASc-score) by either Vitamin-K antagonists (VKAs) or Novel Oral Anticoagulants (NOACs). This allows for a 70% stroke risk reduction.

Not all AF is known to its carrier, it has been proven that 30% of all cases proceeds asymptomatic. These patients are unknowingly exposed to a higher stroke risk. Undertreated AF is when AF is known, but OAC is unrightfully withheld. In approximately 20% of all AF-related strokes, AF was known but undertreated.

In view of the increasing prevalence of AF, it seems there is a need for screening for prevention of actionable AF-associated strokes. The European Society of Cardiology discloses in their most recent guideline that opportunistic screening appears feasible and cost-effective in patients older than 65 years, to be performed by either pulse taking or ECG rhythm strip. The MyDiagnostick, a compact hand-held, 1-lead ECG recorder was created to fulfil the need for better large scale screening devices. In one minute it distinguishes irregular rhythms from normal cardiac rhythms and it can store over 120 ECGs. In a study of 192 patients the MyDiagnostick showed to be 100% sensitive for detecting AF and had a specificity of 95.9%. It provided in a study in which the prevalence of silent AF was examined during influenza vaccination in 10 general practices with more than 3000 patients. From a total of 3269 screened patients, 121 (3,7%) cases of AF were detected, whereof 37 (1,1%) had not yet been diagnosed before.

In this study, the yield of opportunistic screening will be tested of all patients aged 65 or older during preoperative consultation with the MyDiagnostick

ELIGIBILITY:
Inclusion Criteria:

* >64 years of age, visiting preoperative consultation

Exclusion Criteria:

* <64 years of age

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Every patient > 64 years can participate in the trial. Patients who visit the preoperative consultation (e.g. before surgery) will be asked to hold the MyDiagnostick for one minute.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2016-11; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Presence of AF | Single time point (when the patient visits the preoperative consultation hour)
  The MyDiagnostick shows regular or irregular RR-interval

SECONDARY OUTCOMES:
Usage of OAC | Single time point (when the patient visits the preoperative consultation hour)
  Usage of OAC

CONTACTS AND LOCATIONS:
Locations (1):
- Martini Ziekenhuis, Groningen, Netherlands